CLINICAL TRIAL: NCT07164781
Title: Effect of Use of Probiotics on Systemic Infection in Critically Ill Patients: a Double Blind, Randomized, Placebo-controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Doaa kamal Ahmed Ibrahim Qutb, Assistant lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD 10-4-2025
Record Dates: First submitted 2025-05-24; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Acquired Pneumonia; Catheter Related Bloodstream Infection; Urinary Tract Infection; Diarrhea; Probiotics
Keywords: Probiotic; Systemic infection
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Urinary Tract Infections; Diarrhea; Toxemia | interventions — clausin peptide, Bacillus clausii; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The (Control group) will receive placebo (sugar tablets)
  Interventions: Other: Sugar tablets
- Test group (Experimental): The (Test group) will receive bacillus clausii (Enterogermina) 4 billion every 12h.
  Interventions: Biological: Bacillus clausii

INTERVENTIONS:
Biological: Bacillus clausii — The (Test group) will receive bacillus clausii (Enterogermina) 4 billion every 12h.
  Arms: Test group
Other: Sugar tablets — The (Control group) will receive placebo (sugar tablets).
  Arms: Control group

SUMMARY:
The primary goal of this study is to assess the benefit of probiotics in preventing or minimizing of various type of systemic infection in critically ill adult patients.

DETAILED DESCRIPTION:
Healthcare-associated infections constitute a major focus of public health because of their consequences in terms of mortality, morbidity, and financial costs. Owing to multiple pathophysiological factors, such as immune dysfunction or digestive barrier dysfunction, the critically ill patient is indeed particularly prone to Healthcare-associated infections, often after an early colonization of the digestive tube by resistant bacteria. Among these infections, ventilator-associated pneumonia , with an incidence around 15% and an attributable mortality and other Infections such as sepsis, and urinary tract infections remain among the major causes of worsening of the patient's status or even death in critically ill patients.

Ventilator-associated pneumonia is a common pneumonia occurring more than 48 h after endotracheal intubation in the intensive care unit . The duration of mechanical ventilation is positively correlated with the incidence of ventilator-associated pneumonia. ventilator-associated pneumonia has been reported to occur in approximately 40% of patients experiencing mechanical ventilation. By prolonging the duration of mechanical ventilation and intensive care unit stays and increasing antibiotic demands, Ventilator-associated pneumonia usually negatively impacts the Prognosis of critically ill patients.

Central line-associated bloodstream infections are a source of morbidity and impose an important financial burden. As a public safety net health system, we continually strive to improve the quality of our care and to minimize cost. Every health care associated infection is scrutinized to assess whether it could have been prevented. To our surprise, one patient recently fulfilled the National Healthcare Safety Network surveillance definition for a Central line-associated bloodstream infections in a situation which could have been avoided if Probiotics were more carefully handled.

Urinary tract infection is a common bacterial infection that can lead to significant morbidity including stricture, abscess formation, fistula, bacteremia, sepsis, and pyelonephritis and kidney dysfunction. Mortality rates are reported to be as high as 1% in men and 3% in women due to development of pyelonephritis. Because probiotic therapy is readily available without a prescription, a review of their efficacy in the prevention of Urinary tract infection may aid consumers in making informed decisions about potential prophylactic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 18 years or older
* Critically ill patients (medical and surgical) with Acute Physiology and Chronic Health Evaluation II >=10

Exclusion Criteria:

* Patients with active cancer/on chemotherapy and/or radiotherapy/autoimmune diseases/ immunomodulating drugs/ neutropenic fever.
* Pregnancy
* Relatives refuse to share in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of systemic infections | one month

SECONDARY OUTCOMES:
ICU length of stay | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No